CLINICAL TRIAL: NCT06152874
Title: The Combined Effect of Gluten Addition and Cell Wall Integrity in Durum Wheat Bread on Glycemic and Insulinemic Response in Vivo.
Brief Title: Glycemic and Insulinemic Response of Durum Wheat Bread
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Udine (Other)
Collaborators: Wageningen University and Research (Other)
Responsible Party: Principal Investigator, Nicoletta Pelegrini, Professor, University of Udine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: W_D_UDI1
Record Dates: First submitted 2023-10-30; First posted 2023-12-01 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Glucose Response; Glycemic Index; Insulin Response; Oral Processing
Keywords: glucose; insulin; durum wheat bread; oral processing; salivary amylase activity
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- glucose solution 1 (Active Comparator): glucose solution prepared dissolving 55 g of monohydrate glucose powder in 250 mL of water
  Interventions: Other: consumption of glucose solution 1
- glucose solution 2 (Active Comparator): glucose solution prepared dissolving 55 g of monohydrate glucose powder in 250 mL of water
  Interventions: Other: consumption of glucose solution 2
- BREAD A (Experimental): bread made with 95% durum wheat fine semolina (< 400 micrometer)+ 5% of gluten+ 1.2% of yeast + 1% of salt + 59% of water (portion corresponding to 50 g available carbohydrates) +250 mL water
  Interventions: Other: consumption of Bread A and oral processing
- BREAD B (Experimental): bread made with 80% durum wheat fine semolina (< 400 micrometer)+ 20% of gluten+ 1.2% of yeast + 1% of salt + 59% of water (portion corresponding to 50 g available carbohydrates) +250 mL water
  Interventions: Other: consumption of Bread B and oral processing
- BREAD C (Experimental): bread made with 80% durum wheat coarse semolina (> 500 micrometer)+ 20% of gluten+ 1.2% of yeast + 1% of salt + 59% of water) (portion corresponding to 50 g available carbohydrates) +250 mL water
  Interventions: Other: consumption of Bread C and oral processing

INTERVENTIONS:
Other: consumption of glucose solution 1 — glucose solution prepared dissolving 55 g of monohydrate glucose powder in 250 mL of water
  Other Names: glucose solution
  Arms: glucose solution 1
Other: consumption of glucose solution 2 — glucose solution prepared dissolving 55 g of monohydrate glucose powder in 250 mL of water
  Other Names: glucose solution
  Arms: glucose solution 2
Other: consumption of Bread A and oral processing — bread made with 95% durum wheat fine semolina (< 400 micrometer) + 5% of gluten + 1.2% of yeast + 1% of salt + 59%of water) (portion corresponding to 50 g available carbohydrates) + 250 mL water
  Arms: BREAD A
Other: consumption of Bread B and oral processing — bread made with 80% durum wheat fine semolina (< 400micrometer) + 20% of gluten+ 1.2% of yeast + 1% of salt + 59%of water (portion corresponding to 50g available carbohydrates) +250 mL water
  Arms: BREAD B
Other: consumption of Bread C and oral processing — bread made with 80% durum wheat coarse semolina (> 500micrometer)+ 20% of gluten+ 1.2% of yeast + 1% of salt + 59%of water (portion corresponding to 50g available carbohydrates) +250 mL water
  Arms: BREAD C

SUMMARY:
In the last decades, the consumption of energy-dense diets, primarily consisting of highly digestible starchy foods like bread, along with a global increase in obesity rates and a sedentary lifestyle, has emerged as the main contributors to the development of non-communicable diseases such as cardiovascular diseases (CVD) and diabetes type 2. Therefore, there is a need to reduce the starch digestibility of bakery products, and in turn their glycemic index, with a specific emphasis on wheat bread. Several strategies have been used to decrease the glycemic index and insulin response of bread; however, most of these techniques have a detrimental effect on the texture, volume, taste, and color of bread, limiting the consumer's acceptability. Preservation of the native microstructure (cell wall integrity) and employing processing techniques to create a macrostructure (protein network and food matrix) can be used to influence the product structure and therefore how the product is chewed (oral processing), and how these factors can affect carbohydrate digestion and glycemic response. The aim of this study was to examine the effect of different textural characteristics of bread on oral processing in relation to the glycemic and insulin response of the three breads. In the present study, a total of 16 healthy volunteers will be recruited, and if eligible (they need to meet the inclusion and exclusion criteria), they will attend an oral processing test on three breads, a test to measure the glycemic index (ISO) and insulin response.

The bread sample composition will be as follows:

Bread A is made with 95% durum wheat fine semolina (< 400 micrometer) + 5% gluten+ 1.2% yeast + 1% salt + 59% water Bread B is made with 80% durum wheat fine semolina (< 400 micrometer) + 20% gluten+ 1.2% yeast + 1% salt + 59 % water Bread C is made with 80% durum wheat coarse semolina (> 500 micrometer) + 20% gluten+ 1.2% yeast + 1% salt + 59 % water.

DETAILED DESCRIPTION:
Worldwide, the number of people suffering from type 2 diabetes is around 422 million, and this number is continuously rising. It is globally agreed that, by 2025, serious action against the spread of this disease must be taken, also because diabetes is a major cause of the development of cardiovascular diseases. The spread of diabetes in the last decades is the result of a global rise in obesity, a more sedentary lifestyle, and an energy-dense diet, given the overconsumption of mainly highly digestible starchy food. Among highly digestible starchy foods, bread is a staple food consumed daily in western countries and is characterized by a high glycemic index. Carbohydrate-rich foods can be divided into three categories depending on their glycemic index (GI) (low: GI < 55, medium: 55 < GI < 69, or high: GI > 70). This classification is based on how the consumption of food containing carbohydrates affects the blood glucose level in relation to a reference food (such as glucose solution or white bread), which has the same quantity of available carbohydrates (50 g). Foods with a high GI induce a significant rise in postprandial blood glucose concentration and, consequently, a high insulin response, which could lead to hyperinsulinemia and insulin resistance. For this reason, how to decrease the blood glucose response of starchy foods, such as bread, and consequently its GI, has been extensively studied in the last few decades. In plant food, starch granules are naturally encapsulated in the cell. For cereals, the intact cell could limit the accessibility of starch in flours (wheat, sorghum, and barley) and simple food products such as porridge both in vitro and in vivo. However, when coarse flour containing intact cells is used to produce complex foods, such as bread, this effect of protection is lost. The authors hypothesized that during the long mixing time and fermentation, the cell walls increased their porosity due to the solubilization of the cell wall components, such as beta-glucans and arabinoxylans, increasing the diffusivity of the enzymes inside the cell. Moreover, in bread, the addition of coarse flour could also limit the cohesiveness of the crumb, increasing the disintegration rate and, in turn, the contact surface between the enzyme and its substrate. For these reasons, coarse flour could not efficiently decrease the in vitro starch digestibility of bakery products. Protein, the second macronutrient present in cereals, also has a role in decreasing starch digestibility. Gliadin and glutenin, which are the main proteins of wheat grain, formed a discontinuous network that surrounded the starch granules, named gluten. It has been demonstrated that a dense and compact gluten network could decrease starch accessibility, acting as a barrier between starch and enzyme.More specifically, in pasta, its lower glucose release and, in turn, its lower GI compared to bread must be researched in light of the dense and compact structure given by the strong gluten network. Indeed, the dense structure of pasta limits disintegration during oral processing and gastric digestion. This leads to lower postprandial glycemic and insulinemic responses compared to foods with the same recipe but a more porous and easier-to-disintegrate structure. A strong gluten network in bread could, therefore, change the crumb structure, increasing the crumb cohesiveness and resilience.

There is mounting evidence that demonstrates that food structure plays an important role in the digestion and absorption of nutrients. Bread texture affects bread disintegration during the gastric phase, but it mainly influences oral processing and the mastication rate. Oral processing behavior contributes to individual differences in glycemic response to foods, especially in plant tissue, where chewing behavior can modulate the release of starch from the cellular matrix. The addition of gluten cannot only physically hamper the contact between starch and enzyme and reduce the physical disintegration during gastric digestion, but it was also demonstrated that this protein complex could bind pancreatic alpha-amylase and consequently inhibit starch digestibility. The aim of this study is to examine the effect of different textural characteristics of bread on oral processing in relation to the glycemic and insulinemic responses of the three breads. A total of 16 healthy volunteers will be recruited, and if eligible (they need to meet the inclusion and exclusion criteria), they will attend an oral processing test on three breads, a test to measure the glycemic index (ISO) and insulin response.

The bread sample composition will be as follows:

Bread A is made with 95% durum wheat fine semolina (< 400 micrometer) + 5% gluten+ 1.2% yeast + 1% salt + 59% water Bread B is made with 80% durum wheat fine semolina (< 400 micrometer) + 20% gluten+ 1.2% yeast + 1% salt + 59 % water Bread C is made with 80% durum wheat coarse semolina (> 500 micrometer) + 20% gluten+ 1.2% yeast + 1% salt + 59 % water.

For the determination of glycaemic index and insulin response, one fasting capillary blood sample will be taken within 5 minutes, immediately after the participants arrive in the departments. These blood sample results will be used as the baseline blood glucose concentration, expressed in millimoles per liter (mmol/L), and insulin concentration, expressed in milliliters per liter (mU/L). The bread samples and the glucose solution will contain 50 g of available carbohydrates. The different bread samples and glucose solutions will be served to the volunteers using a randomized schedule, and they will finish the portion within 12 to 15 minutes. Test foods will be served with 250 mL of room-temperature natural water; each subject will be asked to drink the same volume for all the tests. The blood sample will be taken at six points (15, 30, 45, 60, 90, and 120 minutes) after the exact time at which the participant started to consume the sample. During testing, the subjects will rest and stay seated. Capillary blood samples will be taken by finger-prick analysis using a sampling lancet (21G x 1.8 mm, ACCU-CHEK Safe-T-Pro Plus, Roche, Switzerland). The blood will be collected in two tubes. At each time point, 3-4 drops of blood will be collected in one Microvette® CB 300 Fluoride/Heparin (SARSTEDT AG & Co., Nümbrech, Germany) for the analysis of capillary blood glucose, and 6-8 drops will be collected in one Microvette® B 300 K2E (Sarstedt Ltd., Germany) for the analysis of plasma insulin. The tubes collected for blood glucose will be immediately analyzed, while plasma from the second set of tubes will be obtained after centrifugation at 4500 rpm for 10 min at 4 °C (Labnet Hermle tabletop Centrifuge Z 200 M/H, Labnet International, Inc., New York, USA) and stored at -80 °C for insulin determination. Blood glucose analysis will be performed using the YSI 2500 Biochemistry Analyzer (Yellow Springs Instrument Company, USA). Insulin concentrations in plasma samples will be determined using a specific immunoassay test kit (Mercodia Insulin ELISA 10-1113-10, Mercodia AB-Uppsala, Sweden). Hunger, satiety, and gastrointestinal symptoms ratings after the test meal consumption will be evaluated with a self-reported questionnaire administered to the volunteers to check subjective feelings of fullness, hunger, and gastrointestinal symptoms at specific time points (before eating, [T0], and after, 30, 60, and 120 min) using a 10 cm visual analog scale. Oral processing parameters will be evaluated for each bread sample through video recording. During this session, the participants will be seated in a chair, and in front of them, there will be a desk with a camera approximately 50 cm from their faces. Participants will be instructed to place the whole sample in the mouth (e.g., a single bite) and to chew naturally until the bolus is ready for swallowing. The oral processing behavior will be described by the following parameters, which will be extracted from video recordings manually: Number of chews and swallows; total eating duration in seconds; chewing rate (number of chews per minute). The food bolus will be evaluated for each bread sample through image analysis to determine particle size distribution and the number of particles present in the bolus, as well as the moisture content, saliva content (grams of saliva per 100 g of bread), and saliva incorporation rate (grams of saliva per minute). For the determination of reducing sugars, the participants will be asked to chew and spit two bites of bread. In the first bolus, HCl will be added to immediately stop the alpha-amylase activity, and then the reducing sugar content will be quantified. For the second one, the reaction will be stopped after 15 minutes, and then the reducing sugars will be measured. The reducing sugars will be anlyzed by the 3,5-dinitrosalicylic acid (DNS) method.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-50 years old;
* Have good general health;
* Have normal smell and taste functions;
* Have a normal body mass index (BMI 18.5-24.9 kg/m2) (based on self-reported weight and height).

Exclusion Criteria:

* Have dental braces or a piercing in or around the mouth (except removable piercings);
* Use medications known to affect glucose tolerance and influence digestion and absorption of nutrients (excluding oral contraceptives) - stable doses of oral contraceptives, acetylsalicylic acid, thyroxin, vitamins, and mineral supplements or drugs to treat hypertension are acceptable.
* Have a known history of diabetes mellitus or the use of antihyperglycemic drugs or insulin to treat diabetes and related conditions;
* Have a major medical or surgical event requiring hospitalization within the preceding 3 months;
* Have any food allergy or intolerance for gluten;
* Being pregnant or lactating (self-reported);
* Use medication that may affect the function of taste, smell, mastication, and salivation;

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-23 (Actual)

PRIMARY OUTCOMES:
Post-prandial glycemic response | Time 2 hours (sampling at 0 -fasting-, 15, 30, 45, 60, 90 and 120 minutes)
  Post-prandial glycemic response (incremental area under the curve)

SECONDARY OUTCOMES:
Maximum peak for glucose | Time 2 hours (sampling at 0 -fasting-, 15, 30, 45, 60, 90 and 120 minutes)
  maximum value of postprandial glucose
Maximum peak for insulin | Time 2 hours (sampling at 0 -fasting-, 15, 30, 45, 60, 90 and 120 minutes)
  maximum value of postprandial insulin
Satiety using a 10 cm Visual Analogue Scale | Time 2 hours (before the meal and after the meal at 30, 60 and 120 minutes)
  Differences in subject-rated satiety using a Visual Analogue Scale consist of a 10 cm line with two endpoints representing 0 ('no satisfied') and 10 ('fully satisfied'). Higher scores mean a better outcome. The incremental area under the curve will be used to check differences over time.
Gastrointestinal symptoms using a questionnaire with symptoms rated using a 10 cm Visual Analogue Scale | Time 2 hours (before the meal and after the meal at 30, 60 and 120 minutes)
  Differences in subject-rated gastrointestinal symptoms using a Visual Analogue Scale consist of a 10 cm line with two endpoints representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). Higher scores mean a worse outcome. The incremental area under the curve will be used to check differences over time.
Post-prandial insulinemic response | Time 2 hours (sampling at 0 -fasting-, 15, 30, 45, 60, 90 and 120 minutes)
  Post-prandial insulinemic response (incremental area under the curve)
Number of chews | Time 5 minutes performed after 2.30 hours of the consumption of samples for the determination of glycemic and insulinemic curves
  The number of chews extracted from the video recorded during bread consumption.
Number of swallows | Time 5 mininutes performed after 2.30 hours of the consumption of samples for the determination of glycemic and insulinemic curves
  The number of swallows extracted from the video recorded during bread consumption
Eating duration | Time 5 minutes performed after 2.30 hours of the consumption of samples for the determination of glycemic and insulinemic curves
  Eating duration extracted from the video recorded during bread consumption
Saliva content in food bolus | Time 5 minutes performed after 2.30 hours of the consumption of samples for the determination of glycemic and insulinemic curves
  The amount of saliva that is incorporated in the food bolus during chewing
Particle size distribution of bolus | Time 5 minutes performed after 2.30 hours of the consumption of samples for the determination of glycemic and insulinemic curves
  The particle size distribution of the bolus, after chewing and spitting in a container, anlyzed with images analysis
Reducing sugar produced in bolus after mastication at time 0 | Time 10 minutes performed after 2.30 hours of the consumption of samples for the determination of glycemic and insulinemic curves
  The amount of reducing sugar produced by alpha-amylase in the bolus immediately after it is spitted in a specific container
Reducing sugar produced in bolus after mastication at time 15 | Time 25 min performed after 2.30 h of the consumption of samples for the determination of glycemic and insulinemic curves
  The amount of reducing sugar produced by alpha-amylase in the bolus after it is spitted in a specific container and incubated for 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Nicoletta Pellegrini, PhD, Principal Investigator — Department of Food Environmental and Animal Sciences
Locations (1):
- Department of Agricultural, Food, Environmental and Animal Sciences, University of Udine,, Udine, Italy

REFERENCES:
- [Background] Tagliasco M, Tecuanhuey M, Reynard R, Zuliani R, Pellegrini N, Capuano E. Monitoring the effect of cell wall integrity in modulating the starch digestibility of durum wheat during different steps of bread making. Food Chem. 2022 Dec 1;396:133678. doi: 10.1016/j.foodchem.2022.133678. Epub 2022 Jul 15. PMID 35849983
- [Background] Vanhatalo S, Dall'Asta M, Cossu M, Chiavaroli L, Francinelli V, Pede GD, Dodi R, Narvainen J, Antonini M, Goldoni M, Holopainen-Mantila U, Cas AD, Bonadonna R, Brighenti F, Poutanen K, Scazzina F. Pasta Structure Affects Mastication, Bolus Properties, and Postprandial Glucose and Insulin Metabolism in Healthy Adults. J Nutr. 2022 Apr;152(4):994-1005. doi: 10.1093/jn/nxab361. Epub 2023 Feb 18. PMID 36967189
- [Background] Dall'Asta M, Dodi R, Pede GD, Marchini M, Spaggiari M, Gallo A, Righetti L, Brighenti F, Galaverna G, Dall'Asta C, Ranieri R, Folloni S, Scazzina F. Postprandial blood glucose and insulin responses to breads formulated with different wheat evolutionary populations (Triticum aestivum L.): A randomized controlled trial on healthy subjects. Nutrition. 2022 Feb;94:111533. doi: 10.1016/j.nut.2021.111533. Epub 2021 Nov 3. PMID 34936948
- [Background] Dhital S, Bhattarai RR, Gorham J, Gidley MJ. Intactness of cell wall structure controls the in vitro digestion of starch in legumes. Food Funct. 2016 Mar;7(3):1367-79. doi: 10.1039/c5fo01104c. PMID 26786854
- [Background] Lau E, Soong YY, Zhou W, Henry J. Can bread processing conditions alter glycaemic response? Food Chem. 2015 Apr 15;173:250-6. doi: 10.1016/j.foodchem.2014.10.040. Epub 2014 Oct 19. PMID 25466020
- [Background] Stamataki NS, Yanni AE, Karathanos VT. Bread making technology influences postprandial glucose response: a review of the clinical evidence. Br J Nutr. 2017 Apr;117(7):1001-1012. doi: 10.1017/S0007114517000770. Epub 2017 May 2. PMID 28462730
- [Background] Zou W, Sissons M, Warren FJ, Gidley MJ, Gilbert RG. Compact structure and proteins of pasta retard in vitro digestive evolution of branched starch molecular structure. Carbohydr Polym. 2016 Nov 5;152:441-449. doi: 10.1016/j.carbpol.2016.06.016. Epub 2016 Jun 3. PMID 27516291
- [Background] Korompokis K , De Brier N , Delcour JA . Differences in endosperm cell wall integrity in wheat (Triticum aestivum L.) milling fractions impact on the way starch responds to gelatinization and pasting treatments and its subsequent enzymatic in vitro digestibility. Food Funct. 2019 Aug 1;10(8):4674-4684. doi: 10.1039/c9fo00947g. Epub 2019 Jul 11. PMID 31292590
- [Background] Chen X, He X, Zhang B, Sun L, Liang Z, Huang Q. Wheat gluten protein inhibits alpha-amylase activity more strongly than a soy protein isolate based on kinetic analysis. Int J Biol Macromol. 2019 May 15;129:433-441. doi: 10.1016/j.ijbiomac.2019.01.215. Epub 2019 Feb 1. PMID 30716375
- [Background] Edwards CH, Grundy MM, Grassby T, Vasilopoulou D, Frost GS, Butterworth PJ, Berry SE, Sanderson J, Ellis PR. Manipulation of starch bioaccessibility in wheat endosperm to regulate starch digestion, postprandial glycemia, insulinemia, and gut hormone responses: a randomized controlled trial in healthy ileostomy participants. Am J Clin Nutr. 2015 Oct;102(4):791-800. doi: 10.3945/ajcn.114.106203. Epub 2015 Sep 2. PMID 26333512
- [Background] Chatterjee S, Khunti K, Davies MJ. Type 2 diabetes. Lancet. 2017 Jun 3;389(10085):2239-2251. doi: 10.1016/S0140-6736(17)30058-2. Epub 2017 Feb 10. PMID 28190580
- [Background] Chen Y, Capuano E, Stieger M. Chew on it: influence of oral processing behaviour on in vitro protein digestion of chicken and soya-based vegetarian chicken. Br J Nutr. 2021 Nov 14;126(9):1408-1419. doi: 10.1017/S0007114520005176. Epub 2020 Dec 28. PMID 33645495
- [Background] Gao J, Lin S, Jin X, Wang Y, Ying J, Dong Z, Zhou W. In vitro digestion of bread: How is it influenced by the bolus characteristics? J Texture Stud. 2019 Jun;50(3):257-268. doi: 10.1111/jtxs.12391. Epub 2019 Feb 14. PMID 30693521
- [Background] Li HT, Li Z, Fox GP, Gidley MJ, Dhital S. Protein-starch matrix plays a key role in enzymic digestion of high-amylose wheat noodle. Food Chem. 2021 Jan 30;336:127719. doi: 10.1016/j.foodchem.2020.127719. Epub 2020 Aug 1. PMID 32768911
- [Background] Mosca AC, Moretton M, Angelino D, Pellegrini N. Effect of presence of gluten and spreads on the oral processing behavior of breads. Food Chem. 2022 Mar 30;373(Pt B):131615. doi: 10.1016/j.foodchem.2021.131615. Epub 2021 Nov 16. PMID 34839974
- [Derived] Tagliasco M, Capuano E, Dall'Asta M, Renzetti S, Fogliano V, Pellegrini N. The combined effect of gluten addition and semolina cell wall integrity reduces the oral sugar release and the insulinemic response to bread in healthy volunteers. Eur J Nutr. 2024 Nov 15;64(1):6. doi: 10.1007/s00394-024-03517-5. PMID 39546030